CLINICAL TRIAL: NCT04889430
Title: A Multicenter, Single-arm, Open Label Trial to Evaluate Efficacy and Safety of Oral, Twice Daily LNP023 in Adult aHUS Patients Who Are Naive to Complement Inhibitor Therapy
Brief Title: Efficacy and Safety of Iptacopan (LNP023) in Adult Patients With Atypical Hemolytic Uremic Syndrome Naive to Complement Inhibitor Therapy
Acronym: APPELHUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023F12301; 2020-005186-13 (EudraCT Number)
Record Dates: First submitted 2021-05-07; First posted 2021-05-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Atypical Hemolytic Uremic Syndrome
Keywords: LNP023; iptacopan; aHUS; atypical hemolytic uremic syndrome; thrombotic microangiopathy
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome; Thrombotic Microangiopathies | interventions — iptacopan

STUDY DESIGN:
Masking Description: Open label single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Iptacopan 200 mg b.i.d (Experimental): Single arm open-label with 50 adult patients receiving 200mg oral twice daily doses of iptacopan
  Interventions: Drug: Iptacopan

INTERVENTIONS:
Drug: Iptacopan — Iptacopan 200mg twice daily oral
  Other Names: LNP023

SUMMARY:
The purpose of this Phase 3 study is to determine whether iptacopan (LNP023) is efficacious and safe for the treatment of aHUS in adult patients who are treatment naive to complement inhibitor therapy.

DETAILED DESCRIPTION:
The study is designed as a multicenter, single-arm, open label study to demonstrate the efficacy and safety of LNP023 (iptacopan) at a dose of 200 mg b.i.d. in adult patients with aHUS who are treatment naive to complement inhibitor therapy (including anti-C5 antibody). The study will enroll approximately 50 participants and assess the effects of iptacopan on a range of efficacy assessments relevant to aHUS including hematological and kidney parameters, dialysis requirement, changes in chronic kidney disease (CKD) stage, as well as patient reported outcomes (PRO) for fatigue and quality of life.

ELIGIBILITY:
Main Inclusion Criteria:

* Adult patients with evidence of active thrombotic microangiopathy (TMA), including thrombocytopenia, evidence of hemolysis, and acute kidney injury
* Vaccinations against Neisseria meningitidis, Streptococcus pneumoniae and Haemophilus influenzae infections are required prior to the start of study treatment. If the patient has not been previously vaccinated, or if a booster is required, vaccine should be given according to local regulations, at least 2 weeks prior to first study drug administration. If study treatment has to start earlier than 2 weeks post vaccination or before vaccination is given, prophylactic antibiotic treatment must be administered at the start of study treatment and for at least 2 weeks after vaccination

Main Exclusion Criteria:

* Treatment with complement inhibitors, including anti-C5 antibody
* ADAMTS13 deficiency (<10% activity or <0.1U/ml), and/or Shiga toxin-related hemolytic uremic syndrome (STx-HUS), and/or Positive direct Coombs test
* Identified drug exposure-related HUS or HUS related to known genetic defects of cobalamin C metabolism or known diacylglycerol kinase ε (DGKE) mediated aHUS
* Receiving PE/PI, for 14 days or longer, prior to the start of screening for the current TMA
* Bone marrow transplantation (BMT)/hematopoietic stem cell transplantation (HSCT), heart, lung, small bowel, pancreas, or liver transplantation
* Patients with sepsis or active severe systemic bacterial, viral (including COVID-19) or fungal infection, systemic infection which confounds an accurate diagnosis of aHUS or impedes the ability to manage the aHUS disease, active infection (or history of recurrent invasive infections) caused by encapsulated bacteria
* Kidney disease suggestive of other disease than aHUS or of chronic kidney failure or family history of non-complement mediated genetic kidney disease
* Liver disease or liver injury at screening
* Systemic sclerosis (scleroderma), systemic lupus erythematosus (SLE), or antiphospholipid antibody positivity or syndrome
* Chronic hemo- or peritoneal dialysis

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2028-09-19 (Estimated); Study Completion 2029-03-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with complete TMA response without the use of PE/PI and anti-C5 antibody | 26 weeks of study treatment
  The number/percentage of participants treated with iptacopan achieving complete thrombotic microangiopathy (TMA) response during 26 weeks of study treatment.
  Complete TMA Response is defined as (1) hematological normalization in platelet count (platelet count ≥150 x 10^9/L) and LDH (below ULN), and (2) improvement in kidney function (≥ 25% serum creatinine reduction from baseline), maintained for two measurements obtained at least four weeks apart, and any measurement in between
Long term safety and efficacy evaluations | 52 weeks of study treatment
  Long term (one year) safety, tolerability and efficacy of iptacopan via 1) safety evaluations including adverse events/serious adverse events, safety laboratory parameters, vital signs etc. after 52 weeks of study treatment, and 2) efficacy evaluations including complete TMA response, hematological parameters (platelets, LDH, hemoglobin), eGFR, PROs after 52 weeks of study treatment

SECONDARY OUTCOMES:
Time to achieve complete TMA response | 26 weeks of study treatment
  Effect of study treatment iptacopan on time to complete TMA response during the first 26 weeks of study treatment
Percentage of participants with increase from baseline in hemoglobin levels ≥ 2 g/dL | 26 weeks of study treatment
  Response is defined as the percentage of participants with an increase in hemoglobin of ≥ 2 g/dL from baseline, observed at two measurements obtained at least 4 weeks apart and any measurement in between during 26 weeks of study treatment
Change from baseline on hematologic parameters | At week 26
  Change from baseline in hematologic parameters (platelets, LDH, hemoglobin) at Week 26
Percentage of participants on dialysis | 26 weeks of study treatment
  For participants requiring dialysis within 5 days prior to iptacopan treatment initiation, the number of participants who no longer require dialysis through 26 weeks of study treatment will be evaluated by means of proportion and corresponding confidence interval
Change from baseline on estimated glomerular filtration rate | At week 26
  Change from baseline in eGFR after 26 weeks of study treatment.
Change from baseline in chronic kidney disease (CKD) stage | At week 26
  Change from baseline in CKD stage (1-5) based on eGFR categories at Week 26
Change from baseline in patient-reported outcomes score as measured by the Functional Assessment Of Chronic Illness Therapy (FACIT)-Fatigue Questionnaire | At week 26
  Change from baseline in patient-reported outcomes scores for FACIT-Fatigue Questionnaire at Week 26
Change from baseline in patient-reported outcomes score as measured by the EuroQol 5-level EQ-5D version (EQ-5D-5L) Questionnaire | At Week 26
  Change from baseline in patient-reported outcomes scores for the EuroQol 5-level EQ-5D version (EQ-5D-5L) Questionnaire at Week 26
Change from baseline in patient-reported outcomes score as measured by the Patient Global Impression of Severity (PGIS) questionnaire | At Week 26
  Change from baseline in patient-reported outcomes scores for Patient Global Impression of Severity (PGIS) at Week 26
Change from baseline in patient-reported outcomes score as measured by the Short-form 36 health survey questionnaire version 2 (SF-36 v2) | At Week 26
  Change from baseline in patient-reported outcomes scores for Short-form 36 health survey questionnaire version 2 (SF-36 v2) at Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- United States (20):
  - Uni Of Alabama At Birmingham, Birmingham, Alabama
  - USC Norris Cancer Center, Los Angeles, California
  - Univ of California at Los Angeles, Los Angeles, California
  - Univ Cali Irvine ALS Neuromuscular, Orange, California
  - Univ of California at Sacramento, Sacramento, California
  - Harbor-UCLA Medical Center ., Torrance, California
  - Georgetown University Lombardi Cancer Center, Washington D.C., District of Columbia
  - University Of Miami, Miami, Florida
  - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - St Barnabas Hospital, Livingston, New Jersey
  - Rut Univ for Translational Med Scie, New Brunswick, New Jersey
  - Montefiore Medical Center ., The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Comprehensive Transplant Ctr at OSU, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Novartis Investigative Site, Vienna, Austria
- Brazil (9):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Recife, Pernambuco
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Botucatu, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, Salvador
- China (6):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Yantai, Shandong
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Ostrava, Poruba, Czechia
- India (8):
  - Novartis Investigative Site, Thiruvananthapuram, Kerala
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Chandigarh, Punjab
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
- Japan (3):
  - Novartis Investigative Site, Iruma-gun, Saitama
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
- Slovakia (2):
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Martin, Slovakia
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Taiwan (2):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient level data and supporting clinical documents from eligible studies. these requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.